CLINICAL TRIAL: NCT06879652
Title: The Effect of Dairy Intake on Body Weight and Composition and Metabolic Health in Adolescents and Seniors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 48001
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-03

CONDITIONS: Dairy Consumption; Metabolic Health; Obesity Prevention
Keywords: Dairy intake; Obesity; Type2 Diabetes; HbA1c; BMI z-score; Insulin resistance; Adolescents; Seniors
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention arm, Dairy Group- Adolescents (Experimental): The participants in the intervention group will consume 3 servings of dairy per day.
  Interventions: Other: Increasing Dairy intake
- Control arm, Low Dairy- Adolescents (No Intervention): The participants in the control group will be asked to maintain their usual diet and dairy intake, involving consuming ≤1 serving of dairy per day.
- Intervention arm, Dairy Group- Seniors (Experimental): The participants in the intervention group will consume 3 servings of dairy per day.
  Interventions: Other: Increasing Dairy intake
- Control arm, Low Dairy- Seniors (No Intervention): The participants in the control group will be asked to maintain their usual diet and dairy intake, involving consuming ≤1 serving of dairy per day.

INTERVENTIONS:
Other: Increasing Dairy intake — The prediabetic and overweight participants aged 14-17 and 60-75 years consuming ≤1 serving of dairy per day who are assigned to the intervention group will consume 3 servings of dairy (milk, yogurt, cheese) before each meal throughout a day for 24 weeks.
  Arms: Intervention arm, Dairy Group- Adolescents; Intervention arm, Dairy Group- Seniors

SUMMARY:
The goal of this study is to examine how regular dairy intake affects body weight, body composition, and metabolic health in overweight and prediabetic adolescents (ages 14-17) and older adults (ages 60-75) over a six-month period. We are inviting eligible individuals to participate in this study at the Nutrition Intervention Center, Department of Nutritional Sciences, University of Toronto, St. George campus. Participants will be randomly divided into two groups. The intervention (high-dairy) group will consume three servings of dairy per day (milk, yogurt, and cheese) before breakfast, lunch, and dinner. The control (low-dairy) group will continue their usual diet, keeping dairy intake less than one serving per day.

Participants will have biweekly sessions with a registered dietitian to monitor their dietary intake and ensure compliance with their assigned group. In addition, they will visit the Nutrition Intervention Center at week 0, week 12, and week 24 for anthropometric and body composition assessments (weight, height, waist circumference, blood pressure, lean mass, fat mass), glycemic and metabolic markers (fasting blood glucose, insulin, HbA1c, lipid profiles in seniors, and appetite hormones in adolescents). Each assessment visit will take approximately 4 hours.

Before each visit, you will be asked to fast for 12 hours overnight, maintain your usual diet and sleep patterns, and avoid exercise and alcohol consumption the day before. Your participation in this study will help us better understand the role of dairy in metabolic health and may contribute to improved dietary recommendations for adolescents and older adults. You will be compensated for your time and travel expenses.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-17 years old (adolescents) or 60-75 years old (seniors)
* BMI z-score >+1SD, <+2SD (adolescents) or BMI 25-30 kg/m2 (seniors)
* Waist circumference > 88 cm for women and > 102 cm for men (seniors)
* FBG 5.6-6.9 mmol/L (prediabetes)
* Consumes ≤1 serving of dairy per day
* Willing to maintain habitual diet, physical activity, and body weight throughout the study.
* Willing to maintain current dietary supplement use throughout the study. On the first day, the participants agree not to take any dietary supplements until the completion of the study.
* Willing to abstain from alcohol consumption for 24 hours prior to all test visits.
* Willing to avoid vigorous physical activity for 24 hours prior to all test visits.
* Understands the study procedures and is willing to provide informed consent by parent/guardian and assent by participant to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Fasting BG ≥ 7mmol/L
* Blood pressure systolic ≥ 130mmHg or diastolic ≥ 80mmHg (adolescents) or systolic ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg
* Smoking (tobacco and/or cannabis product use in the last 6 months)
* Thyroid problems
* History of CVDs, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorption syndrome, pancreatitis, gallbladder, or biliary disease.
* Presence of gastrointestinal disorder or surgeries within the past year.
* Use of the prescription or non-prescription drugs, herbal or nutritional supplements known to affect the outcome of the study as per the investigator's judgment (including prebiotics and probiotics).
* History of childhood obesity
* Known to be pregnant, lactating, or not postmenopausal for at least a year and/or is taking hormonal treatments
* Unwillingness or inability to comply with the experimental procedures
* Known intolerance, sensitivity, or allergy to dairy, gluten, or any other study treatments.
* Consumption of protein powders/supplements
* Extreme dietary habits (e.g., Atkins diet, very high-protein diets, etc.)
* Weight gain or loss of >10 lbs. in the previous three months.
* Excessive alcohol intake (more than 2 drinks per day or 9 per week)
* Restrained eating, identified by a score of ≥11 on the Eating Habits Questionnaire

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c (%) | HbA1c will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  HbA1c measures average blood glucose levels over the past 2-3 months. It will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast.
Body Mass Index (BMI) z-score | BMI z-score will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  BMI z-score is an age- and sex-adjusted measure of BMI in adolescents. It will be calculated using height and weight measurements and interpreted using WHO or CDC growth charts and percentiles.

SECONDARY OUTCOMES:
Fasting blood glucose (FBG) (mmol/L) | FBS will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  FBS will be measured to assess glycemic control. It will be measured using a fingerprick blood sample and a glucometer after a 12-hour overnight fast.
Oral Glucose Tolerance Test (OGTT) (mmol/L) | OGTT will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  OGTT assesses glucose tolerance and insulin response by measuring blood glucose at 0, 15, 30, 45, 60, 90, and 120 minutes after consuming a 75-gram glucose drink using a fingerprick blood sample and a glucometer.
Insulin (µU/mL) | Insulin will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  Insulin levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast.
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | HOMA-IR will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  HOMA-IR will be calculated as (Fasting Insulin [µU/mL] × Fasting Glucose [mmol/L]) / 22.5 to assess insulin resistance.
C-Reactive protein (CRP) (mg/L) | CRP will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  CRP, a marker for assessing systemic inflammation, will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast.
Total cholesterol (TC) (mmol/L) | TC will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  TC levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess lipid metabolism and cardiovascular risk in seniors.
Low-density lipoprotein cholesterol (LDL-C) (mmol/L) | LDL-C will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  LDL-C levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess cardiovascular risk and lipid metabolism in seniors.
High-density lipoprotein cholesterol (HDL-C) (mmol/L) | HDL-C will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  HDL-C levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess cardiovascular health and lipid metabolism in seniors.
Triglycerides (mmol/L) | Triglycerides will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  Triglyceride levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess lipid metabolism and cardiovascular risk in seniors.
C-Peptide (pmol/L) | C-Peptide will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  C-peptide levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess pancreatic beta-cell function and insulin secretion in adolescents.
Glucagon-Like Peptide-1 (GLP-1) (pmol/L) | GLP-1 will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  GLP-1 levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess incretin hormone response and its role in glucose metabolism in adolescents.
Ghrelin (pmol/L) | Ghrelin will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  Ghrelin levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess hunger regulation and appetite control in adolescents.
Peptide YY (PYY) (pmol/L) | PYY will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  PYY levels will be measured in plasma obtained through intravenous blood collection after a 12-hour overnight fast to assess appetite regulation and satiety control in adolescents.
Blood pressure (BP) (mmHg) | BP will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  Blood pressure will be measured using an automated sphygmomanometer after the participant has been seated and at rest for at least 5 minutes. Measurements will include systolic and diastolic blood pressure.
Waist circumference (WC) (cm) | WC will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  WC will be measured to assess abdominal adiposity using a standardized measuring tape at the midpoint between the lowest rib and the iliac crest while the participant is in a standing position.
Body Fat Mass (BFM) (kg) | BFM will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  BFM will be measured using bioelectrical impedance analysis (BIA) and air displacement plethysmography (ADP).
Lean body mass (LBM) (Kg) | LBM will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  LBM will be measured using bioelectrical impedance analysis (BIA) and air displacement plethysmography (ADP)
Body Mass Index (BMI) (kg/m²) | BMI will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  BMI will be calculated to assess overall adiposity in seniors using weight and height measurements, applying the formula: BMI = weight (kg) / height (m²).

OTHER OUTCOMES:
Dietary intake (Kcal, gram) | Dietary intake will be assessed at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  Dietary intake will be assessed using a food frequency questionnaire (FFQ) and a 3-day food record to evaluate energy and macronutrient intake, as well as adherence to the assigned group.
Resting Metabolic Rate (RMR) (kcal/day) | RMR will be measured at the beginning (week 0), midpoint (week 12), and end of the study (week 24).
  RMR will be measured using indirect calorimetry after an overnight fast and at least 30 minutes of rest in a thermoneutral environment.

CONTACTS AND LOCATIONS:
Overall Officials: G Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Department of Nutritional Sciences, Toronto, Ontario
  - Nutrition Intervention Center, Toronto

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, as all data will be de-identified and pooled during the analysis. Only researchers directly involved in the study will have access to the data.